CLINICAL TRIAL: NCT04575961
Title: Phase II Investigational Study of Pembrolizumab Combination With Chemotherapy in Platinum-sensitive Recurrent Low-grade Serous Ovarian Cancer
Brief Title: Study of Pembrolizumab Combination With Chemotherapy in Platinum-sensitive Recurrent Low-grade Serous Ovarian Cancer
Acronym: PERCEPTION
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: North Eastern German Society of Gynaecological Oncology (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOGGO-ov44
Record Dates: First submitted 2020-09-07; First posted 2020-10-05 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-11

CONDITIONS: Ovarian Cancer; Low Grade Serous Carcinoma; Primary Peritoneal Carcinoma; Fallopian Tube Cancer
Keywords: Pembrolizumab; Chemotherapy; Platinum-Sensitive
MeSH Terms: conditions — Ovarian Neoplasms; Cystadenocarcinoma, Serous; Fallopian Tube Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab + Chemotherapie (Other): pembrolizumab in combination with platinum-based chemotherapy (investigator's choice: carboplatin + gemcitabine or carboplatin + pegylated liposomal doxorubicin)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Participants receive pembrolizumab 200 mg by intravenous (IV) infusion prior to chemotherapy on Day 1 of each 21-day cycle for up to 35 cycles
  Other Names: Keytruda

SUMMARY:
This is a phase II, single arm, multi-centre study to assess the efficacy of pembrolizumab in combination with platinum-based chemotherapy (investigator's choice: carboplatin + gemcitabine or carboplatin + pegylated liposomal doxorubicin) administered concurrent to chemotherapy and in maintenance, in patients with low grade ovarian cancer (including patients with primary peritoneal and / or fallopian tube adenocarcinoma) having platinum-sensitive relapse (platinum-free interval > 6 months).

DETAILED DESCRIPTION:
In this study, we will evaluate efficacy and safety of pembrolizumab in combination with chemotherapy (physician's choice) in subjects with low-grade ovarian cancer.

Patients will receive Pembrolizumab 200mg q3w until progression or unacceptable toxicity, for a maximum of 35 cycles PLUS one of the following standard chemotherapies for LGSOC (investigators' choice):

Carboplatin AUC 4 + Gemcitabine 1000mg/m² (q3w for 3-6 cycles) or Carboplatin AUC 5 + pegylated liposomal Doxorubicin 30mg/m² (q4w for 3-6 cycles). As primary objective 12-month progression free survival (PFS) rate will be analysed.

About 2 sites in Germany will participate in this study to recruit 33 patients in 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Female, age at least 18 years.
* Histologically diagnosed low-grade serous ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.
* Patients must have completed at least 1 previous course of platinum-containing therapy (e.g., combination with carboplatin or cisplatin. Maintenance therapy with bevacizumab and/or endocrine agents is allowed).
* Progression or recurrence after platinum-containing therapy, occurring no sooner than 6 months after completion of the last dose of platinum chemotherapy (platinum sensitive disease).
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Women of childbearing potential should not become pregnant while on the Product and should not be pregnant at the beginning of treatment. A pregnancy test should be performed on all women of childbearing potential prior to receiving the Product. Women of childbearing potential must agree to follow contraceptive guidance during the treatment period and for 6 months after receiving the last dose of the study therapy.
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
* Availability of archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.

Exclusion Criteria:

* High-grade ovarian cancer.
* Persistent ≥Grade 2 hematologic toxicity from prior cancer therapy Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.

Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.

* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137).
* Is eligible for carboplatin-based doublet therapy in combination with bevacizumab in the relapse situation, since no treatment with bevacizumab has been administered in the first line therapy.
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks.
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Has a bleeding tumor
* Has hypersensitivity to any of the study drugs the patient will be treated with and/or to any of the excipients of the study drugs the patient will be treated with.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] has been detected) infection.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has had an allogenic tissue/ solid organ transplant.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive within the projected duration of the study, starting with the screening visit through 6 months after the last dose of trial treatment.
* Patients unable to be regularly followed for any reason (geographic, familiar, social, psychologic, housed in an institution e.g. prison because of a court agreement or administrative order).
* Subjects that are depending on the sponsor/CRO or investigational site as well as on the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only women can get ovarian cancer
Enrollment: 33 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
12-month (48 weeks) progression free survival (PFS) rate | 12 month
  The primary objective of this clinical trial is 12-month Progression Free Survival (PFS) rate after start of treatment. Tumor progression will be assessed with local imaging per irRECIST 1.1 and is defined according to RECIST criteria. Start of therapy will be counted when the patient receives the first dose of pembrolizumab.

SECONDARY OUTCOMES:
Response rate (SD, PR or CR) after 6, 12, 18 and 24 months | 6, 12, 18 and 24 months
  Stable Disease, Partial Response or CR will be evaluated per irRECIST 1.1 after 6, 12,18 and 24 months
Ki-67 | 24 month
  Marker of proliferation Ki-67 Obtain archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated for routine determination of PD-1, PD-L1 and Ki-67 status
Time of next medical intervention | 24 month
  Time of next medical intervention due to tumor progress
Quality of life until 6 months after progress | 6 month
  Patients are asked to answer the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30). Responses of questions 1-28 are based on a 4-point scale (1=not at all; 4=Very much), with a higher score indicating a high degree of symptomatology and must therefore be assessed negatively. Responses of questions 29 and 30 are based on a 7-point scale (1=Very poor; 7=Excellent), with a higher score indicating a better global health status.
TFST and response to first subsequent treatment | 24 month
  Time to first subsequent treatment and response to first subsequent treatment will be evaluated.
Safety Endpoints - safety of combination therapy (ctx and pembrolizumab) according to CTCAE 5.0 criteria will be used as endpoint | 24 month
  The safety objective is to characterize the safety and tolerability of pembrolizumab in combination with chemotherapy in subjects with advanced low grade ovarian cancer. The following safety parameters will be analyzed: adverse events and serious adverse events graded per NCI CTCAE, Version 4.0 criteria with time to onset/recovery, causality and outcome; changes in laboratory values, vital signs since baseline, treatment discontinuations and reason for discontinuation, death and cause of death etc. concomitant medications will be collected with time and reasons of use. These are routine safety parameters collected and analyzed in Phase II /III oncology trials. Furthermore, specific immune-related adverse events (irAEs) will be collected
PFS (time-to-event) and PFS rate after 6, 12, 18 and 24 months | 6, 12, 18 and 24 months
  Progression Free Survival (time to event) and PFS rate after 6, 12, 18 and 24 months after start of treatment. Tumor progression will be assessed with local imaging per irRECIST 1.1 and is defined according to RECIST criteria. Start of therapy will be counted when the patient receives the first dose of pembrolizumab
Quality of life 2 until 6 months after progress | 6 month
  Patients are asked to answer the EORTC QoL Questionnaire-Ovarian Cancer (QLQ-OV28). Responses are based on a 4-point scale (1=Not at all; 4=Very much), with a lower score indicating better symptoms.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Campus Virchow Klinikum, Berlin
  - Kliniken Essen Mitte, Essen

IPD SHARING:
Plan to Share IPD: Yes
Sciences may submit a request for scientific use of the data after the first publication. This request shall be examined by the working group. After signing an agreement, the anonymous data can be made available to the scientist (password protected).
Supporting Information: Study Protocol, ICF
Time Frame: after first main publication